CLINICAL TRIAL: NCT00979953
Title: A Phase 2a, Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Multicenter Study Evaluating the Analgesic Efficacy and Safety of ADL5859 and ADL5747 in Subjects With Moderate to Severe Pain Due to Osteoarthritis of the Knee
Brief Title: Efficacy and Safety Study Evaluating ADL5859 and ADL5747 in Participants With Pain Due to Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44CL240
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: delta opioid receptor agonist; osteoarthritis; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — N,N-diethyl-4-(5-hydroxyspiro(chromene-2,4'-piperidine)-4-yl)benzamide; N,N-diethyl-3-hydroxy-4-(spiro(chromene-2,4'-piperidine)-4-yl)benzamide; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADL5859 (Experimental): One 50-milligrams (mg) ADL5859 capsule, one 100-mg ADL5859 capsule, and 2 placebo capsules administered orally twice daily (BID) for 14 days
  Interventions: Drug: ADL5859; Drug: Placebo
- ADL5747 (Experimental): One 150-mg ADL5747 capsule and 3 placebo capsules administered orally BID for 14 days
  Interventions: Drug: ADL5747; Drug: Placebo
- Oxycodone CR (Active Comparator): One 10-mg Oxycodone controlled release (CR) capsule and 3 placebo capsules administered orally BID Days 1 through 4
  One 20-mg Oxycodone CR capsule and 3 placebo capsules administered orally BID Days 5 through 14
  Interventions: Drug: Oxycodone CR; Drug: Placebo
- Placebo (Placebo Comparator): Four placebo capsules administered orally BID for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADL5859
  Arms: ADL5859
Drug: ADL5747
  Arms: ADL5747
Drug: Oxycodone CR
  Other Names: OxyContin
  Arms: Oxycodone CR
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of ADL5859 versus placebo and ADL5747 versus placebo in relieving pain in participants with osteoarthritis of the knee.

ELIGIBILITY:
Key Inclusion Criteria:

* a man or woman between 18 and 75 years of age, inclusive
* for women of childbearing potential, be using an insertable, injectable, transdermal, or combination oral contraceptive deemed highly effective by the United States Food and Drug Administration from the first dose of study medication through the end of the study and have negative findings on pregnancy tests performed at screening and randomization (women who are surgically sterile [for example, hysterectomy, tubal ligation] or postmenopausal [if ≥55 years old, no menses for at least 2 years; if <55 years old, follicle-stimulating hormone concentrations within the postmenopausal range of >40 milli-international units per milliliter (mIU/mL) and 17 β-estradiol levels of <37 picograms per milliliter (pg/mL)] are also eligible to participate)
* for male participants, be surgically sterile or agree to use an appropriate method of contraception (that is, use a barrier method in conjunction with spermicide or have a sexual partner who is surgically sterile, postmenopausal, or using an insertable, injectable, transdermal, or combination oral contraceptive deemed highly effective by the United States Food and Drug Administration) from the first dose of study medication through the end of the study
* have a body weight between 45 and 150 kilograms (kg), inclusive
* have had pain in the index knee for at least the past 6 months
* meet the following criteria for osteoarthritis of the knee established by the American College of Rheumatology (radiographs must have been taken within the last year; if none is available, a radiograph must be taken and the diagnostic criteria must be confirmed before the participant is enrolled in the study): have index knee pain plus at least 1 moderate or definite osteophyte on radiographs. Must also have at least 1 of the following: be more than 50 years old, have morning stiffness for less than 30 minutes, or have crepitus on active motion
* have an average weekly pain score of at least 4.00 on the numeric pain rating scale (NPRS) for the index knee during the baseline week before randomization (to be eligible for randomization, participants must report their NPRS score via the interactive voice-response system (IVRS) for at least 4 of the 7 days immediately before randomization, with the first score being recorded on Day -6)
* if receiving nonselective or selective cyclooxygenase (COX) inhibitors, have a stable daily dose regimen for at least 4 weeks before screening; if receiving nonselective or selective COX inhibitors on an as needed basis, have discontinued use by Day -14; if receiving angiotensin-converting enzyme (ACE) inhibitors, have a stable dose regimen for at least 4 weeks before screening

Key Exclusion Criteria:

* have undergone arthroscopy on the index knee within 6 months before study entry
* have other severe pain that, in the opinion of the investigator, may impair the assessment of the pain due to osteoarthritis
* have a history of hypersensitivity or intolerance to opioids (including tramadol and tapentadol)
* have, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant renal, hepatic, hematologic, cardiovascular, metabolic, gastrointestinal, neurologic, psychiatric, or another condition that would preclude participation in the study or affect the outcome of the study
* have taken oral or intramuscular corticosteroids within 30 days before study entry (inhaled or topical corticosteroids are permitted)
* have received intra-articular injections of corticosteroids into the index joint within 12 weeks before screening
* have received intra-articular injections of hyaluronic acid into the index joint within 24 weeks before screening
* currently taking medications other than nonsteroidal anti-inflammatory drugs prescribed for chronic pain (such as duloxetine or pregabalin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Berger, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (11):
- United States (11):
  - Covance CRU, Inc, Daytona Beach, Florida
  - Atlanta Knee and Shoulder Clinic, PC, Stockbridge, Georgia
  - University Rheumatoloty Center for Clinical Research, Chicago, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Cresent Medical Research, Salisbury, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Columbus Clinical Research, Columbus, Ohio
  - PSB Research, Mount Gilead, Ohio
  - Bone Joint & Spine Surgeons, Inc, Toledo, Ohio
  - Radient Research, Anderson, South Carolina
  - Quality Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADL5859 | ADL5747 | Oxycodone CR | Placebo
Started | 101 | 99 | 104 | 104
Received at Least 1 Dose of Study Drug | 101 | 99 | 104 | 104
Completed | 93 | 94 | 82 | 97
Not Completed | 8 | 5 | 22 | 7
Not completed — Adverse Event | 5 | 2 | 17 | 4
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants received at least 1 dose of study drug.
Groups:
- ADL5859: One 50-mg ADL5859 capsule, one 100-mg ADL5859 capsule, and 2 placebo capsules administered orally BID for 14 days
- Oxycodone CR: One 10-mg Oxycodone CR capsule and 3 placebo capsules administered orally BID Days 1 through 4
  One 20-mg Oxycodone CR capsule and 3 placebo capsules administered orally BID Days 5 through 14
- Total: Total of all reporting groups
Arm/Group | ADL5859 | ADL5747 | Oxycodone CR | Placebo | Total
Number analyzed (Participants) | 101 | 99 | 104 | 104 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.15) | 57.3 (8.74) | 57.8 (8.39) | 56.5 (8.11) | 57.0 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 57 | 63 | 61 | 240
  Male | 42 | 42 | 41 | 43 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Pain Score (NPRS) for Week 2
Description: The mean of the daily average scores were calculated from the NPRS pain assessment for the previous 24 hours obtained once a day for at least 4 days from Day -6 through Day 1 (Baseline assessment) and everyday from Day 2 through Day 15 (Treatment Phase assessment). The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain.
Time Frame: Baseline, Week 2
Population: All participants who received at least 1 dose of study medication and had at least evaluable 1 NPRS postdose measurement. Last-observation-carried-forward (LOCF) was used to impute missing postbaseline values.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- Oxycodone CR: One 10-mg Oxycodone CR capsule and 3 placebo capsules administered orally BID Days 1 through 4
  One 20-mg Oxycodone CR capsule and 3 placebo capsules administered orally BID for Days 5 through 14
Arm/Group | Placebo | Oxycodone CR | ADL5747 | ADL5859
Number analyzed (Participants) | 103 | 100 | 99 | 101
units on a scale | -2.20 (2.088) | -2.24 (2.162) | -1.57 (1.656) | -1.77 (1.776)

ADVERSE EVENTS:
Arm/Group | ADL5859 | ADL5747 | Oxycodone CR | Placebo
Serious Adverse Events (participants affected / at risk) | 2/101 | 1/99 | 0/104 | 1/104
Other Adverse Events (participants affected / at risk) | 50/101 | 40/99 | 75/104 | 37/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADL5859 (N=101) | ADL5747 (N=99) | Oxycodone CR (N=104) | Placebo (N=104)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADL5859 (N=101) | ADL5747 (N=99) | Oxycodone CR (N=104) | Placebo (N=104)
Constipation (Gastrointestinal disorders) | 8 | 5 | 30 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 7 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 8 | 6 | 13 | 6
Nausea (Gastrointestinal disorders) | 5 | 5 | 32 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 15 | 0
Fatigue (General disorders) | 6 | 2 | 17 | 7
Dizziness (Nervous system disorders) | 4 | 1 | 17 | 2
Headache (Nervous system disorders) | 10 | 10 | 13 | 3
Somnolence (Nervous system disorders) | 7 | 4 | 20 | 8
Disturbance in attention (Psychiatric disorders) | 2 | 0 | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 17 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other